# Requirements for Submitting a Full Proposal

### Section #1 - MISP Protocol Identification

| Study Title: | An Open-label Pharmacokinetic Study of Imipenem-Cilastatin-Relebactam in Critically-III Patients with Augmented Renal Clearance |
|---|---|
| Request Date: | Original Submission: February 7, 2019 Amendment 1 Version: May 14, 2020 Amendment 2 Version: July 31, 2020 Amendment 3 Version: December 22, 2020 |
| Institution Name | Hartford Hospital |
| Investigator Contact Information: - Full address - Phone No Fax No e-mail address | Joseph L. Kuti, PharmD, FIDP Center for Anti-Infective Research and Development Hartford Hospital 80 Seymour Street Hartford, CT 06102 Tel: 860-972-3612 Fax: 860-545-3992 Email: joseph.kuti@hhchealth.org |

MISP Template: Protocol Final Version: 8/13/2010

IRB NUMBER: HHC-2019-0237
IRB APPROVAL DATE: 12/22/2020

### Section #2- Core Protocol

### 1.0 Amendment 1 – Dated May 14, 2020

- Imipenem-relebactam changed to imipenem-cilastatin-relebactam throughout the protocol to document inclusion of cilastatin. This maintains consistency with the package insert for the drug and also clarifies the dosage.
- 2. The dosage has been changed to 1.25 grams throughout the protocol. This total dose is consistent with the package insert and contains 500mg of imipenem, 500mg of cilastatin, and 250mg of relebactam. Note, the total amount of imipenem and relebactam administered to the patient is not different from the original protocol.
- 3. Section 2.1: correct misspelling
- 4. Section 2.2: Background updated to indicate approval of imipenemcilastatin-relebactam for complicated urinary tract and intra-abdominal infections.
- 5. Section 2.5 modified to indicate collection of blood in K2EDTA lavender tubes instead of sodium heparin tubes. The assay to be used requires K2EDTA tubes for collection. As a result, the maximum blood volume per sample has been reduced from 7 mL to 4 mL, since the latter is the maximum volume of a lavender top tube. Additional details provided on processing of plasma with MES stabilizer.
- 6. Section 2.5 modified to add free drug assessments of imipenem and relebactam.
- Section 2.7 modified to provide details of analytical service by Q2 Solutions, Ithaca NY.
- 8. Section 2.7 modified to incorporate fraction unbound estimates into Monte Carlo simulations.

### 1.1 Amendment 2 – Dated July 31, 2020

1. Section 2.5 modified to indicate collection of additional pre-dose blood sample within 30 minutes of infusion start time.

### 1.2 Amendment 3 – Dated December 22, 2020

- Section 2.5 inclusion criteria #3 modified to lower creatinine clearance (CrCL) from 150 mL/min to 130 mL/min. This has been changed throughout protocol accordingly. This will increase the target population while still limiting patients to those with augmented renal clearance.
- Section 2.5 inclusion criteria #4 modified to include only antibiotic use as a
  method for determining whether or not a patient has a documented or
  presumed infection, and removing other criteria related to infection
  (temperature, elevated WBC).
- 3. Section 2.5 inclusion criteria #10 modified to reduce minimum APACHE II score from >12 to ≥10. The threshold of 12 was arbitrary, while the intent is to include relatively sick patients in the study, which will still be the case.
- 4. Section 2.5 exclusion criteria #9 modified to remove valproic acid.
- Section 2.5 addition of criteria #10 excluding patients currently receiving or anticipated to receive valproic acid. The change in criteria 9 and 10 will allow for patients to receive imipenem-cilastatin-relebactam despite a prior recent history of valproic acid use.

# 2.1 Objectives & Hypotheses

MISP Template: Protocol 2 Final Version: 8/13/2010

### 2.1 Objectives

- 1. Determine the single-dose pharmacokinetics of intravenous imipenem (when administered as imipenem-cilastatin-relebactam 1.25 grams as a 30 minute infusion) in adult critically ill patients with known or suspected sepsis and ARC
- Determine the single-dose pharmacokinetics of intravenous relebactam (when administered as imipenem-cilastatin-relebactam 1.25 grams as a 30 minute infusion) in adult critically ill patients with known or suspected sepsis
- Determine a dose of imipenem-cilastatin-relebactam that achieves greater than 90% probability of pharmacodynamic target attainment using the imipenem P. aeruginosa susceptibility breakpoint of 2 µg/mL and the MIC distribution of a contemporary P. aeruginosa and KPC producing K. pneumoniae population
- 4. Assess the safety and tolerability of single-dose imipenem-cilastatinrelebactam in adult critically ill patients with known or suspected sepsis and **ARC**

### 2.1.1 Null Hypotheses

The pharmacokinetics of imipenem and relebactam will not be affected by the presence of augmented renal clearance in adult critically ill patients.

The continuous rise of bacterial resistance to antibiotics is among the most challenging concerns in contemporary clinical medicine. Imipenem-relebactam (Merck&Co. Inc., Kenilworth, NJ) is an investigational broad-spectrum antibiotic that combines the known carbapenem, imipenem, with the novel beta-lactamase inhibitor, relebactam (1). The addition of relebactam provides imipenem protection against serine based carbapenemases, including the Klebsiella pneumoniae carbapenemase (KPC), as well as improved activity against imipenem nonsusceptible Pseudomonas aeruginosa (2). Imipenem-cilastatin-relebactam is approved in the United States for complicated urinary tract infections and complicated intra-abdominal infections; it is under investigation for hospital-acquired and ventilator-associated pneumonia, and specifically for multidrug resistant Gramnegative infections when it retains activity (1).

2.2 Background & Rationale. Significance of Selected Topic & Preliminary Data

Given its potent activity against KPC producing Enterobacteriaceae and imipenem non-susceptible P. aeruginosa, it is reasonable to consider that imipenemcilastatin-relebactam will be used in patients who are critically ill in the intensive care unit (ICU). Critically ill patients may have varied kidney dysfunction as a result of acute infection. Most clinicians are familiar with acute and chronic kidney impairment, which results in decreased elimination of drugs that are cleared by glomerular filtration. Both imipenem and relebactam are predominantly excreted via the kidneys (3); therefore, dosage adjustments will be required based on calculated creatinine clearance. Sepsis in ICU patients, however, may also produce a syndrome called Augmented Renal Clearance (ARC), whereby increased blood flow to the kidneys results in enhanced renal elimination and solute clearance (4). This enhanced clearance is typically defined by an 8 hour urine creatinine clearance ≥ 130 ml/min/1.73 m<sup>2</sup> and has been observed in as many as 65% of ICU patients on at least one day during their ICU admission (4,5). ARC has been directly linked to subtherapeutic concentrations of β-lactam antibiotics, including imipenem (6,7,8,9). Furthermore, simulation of another carbapenem, meropenem, based on pharmacokinetics observed in patients with ARC resulted in regrowth of a susceptible *Pseudomonas aeruginosa* in hollow-fiber experiments (10).

MISP Template: Protocol 3 Final Version: 8/13/2010

| | To our knowledge, the pharmacokinetics of relebactam, with or without imipenem, have not been studied in critically ill patients with ARC. If ARC affects relebactam clearance to a similar degree as imipenem and other renally eliminated β-lactams, larger doses or prolonged infusion may be required to maintain optimized pharmacodynamic exposure. Importantly, the effect of ARC on beta-lactam exposure is highly dependent on the MIC of the causative organism. Therefore, it is also possible that the lower MICs observed with imipenem when combined with relebactam may mean that ARC has little effect on achievable time above the MIC exposure. |
|---|---|
| 2.3 Study Design | This will be a single center, observational, pharmacokinetic study. Eligible patients will be evaluated for inclusion/exclusion criteria. Following consent by the patient, legal authorized representative (LAR), or next of kin, participants will receive a single dose of imipenem-cilastatin-relebactam 1.25 grams administered as a 30 minute infusion. Blood samples will be collected over the following 6 hours (consistent with proposed dosing interval) for characterization of imipenem and relebactam concentrations. Pharmacokinetic analyses will be conducted to describe parameter estimates in patients with ARC. We aim to enroll up to 12 patients so that complete data for 8 patients with ARC can be collected. |
| 2.4 Study Flowchart | N/A |
| 2.5 Study<br>Procedures | The Center for Anti-Infective Research and Development (CAIRD), Hartford Hospital, CT will coordinate the study. The study will conducted in the medical, surgical, and neurosurgical ICUs at Hartford Hospital, an 890 bed tertiary care hospital in Hartford, CT. Institutional Review Board approval will be required based on local regulations. If LAR or next of kin are consented, local regulations will be followed to collect written informed consent from the patient once able to provide consent. Study Population Inclusion Criteria Patients eligible to participate in the study must meet all of the following criteria prior to any study-related procedure: 1. Male or female aged 18-54 years; 2. APACHE II score ≥ 10 and ≤ 35; 3. Creatinine clearance (CrCL) ≥130 mL/min (as calculated by the Cockcroft-Gault equation using ideal or adjusted body weight) within 24 hours of dosing (Note: using a higher CrCL threshold for Cockcroft-Gault CrCL will increase likelihood that enrolled participants have a urine CrCL ≥ 130 ml/min/1.73 m² and thus qualify as ARC); 4. Documented infection or presumed infection by receiving another antibiotic. Exclusion Criteria Patients will be considered ineligible if they meet any of the following criteria: 1. If female, currently pregnant or breast feeding; 2. History of any moderate or severe hypersensitivity or allergic reaction to any |
| | <ul> <li>β-lactam antibiotic (<i>Note:</i> mild rash or erythema to penicillin or cephalosporin antibiotics would not disqualify a patient if they have received a carbapenem without problem);</li> <li>History of chronic kidney disease, hemodialysis, or peritoneal dialysis; or history of acute renal replacement therapy (e.g., hemodialysis,</li> </ul> |

MISP Template: Protocol 4 Final Version: 8/13/2010

- hemofiltration, hemodiafiltration) or extracorporeal membrane oxygenation (ECMO) associated with current illness:
- 4. Suspected rhabdomyolysis or creatine kinase > 10,000 U/L;
- 5. Any serum creatinine (SCr) before dosing that is increased ≥ 0.3 mg/dL from the baseline SCr used qualifying for enrollment:
- 6. Urinary output <20 ml/hour for at least 2 hours (oliguria) within 24 hours before enrollment:
- 7. Sustained (at least 1 hour) hypotension (systolic pressure < 90 mmHG or mean arterial pressure < 55 mmHg) refractory to vasopressors or IV fluid resuscitation for at least 24 hours before enrollment;
- Significant anemia defined as a hemoglobin < 8 g/dL at baseline;
- Use of probenecid or imipenem within 3 days before study drug infusion:
- 10. Current use of valproic acid or anticipated use during study enrollment.
- 11. Acute liver injury, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 times the upper limit of normal, or AST or ALT > 3 times the upper limit of normal with an associated total bilirubin > 2 times upper limit of normal;
- 12. Any rapidly-progressing disease or immediately life-threatening illness (defined as imminent death within 48 hours in the opinion of the investigator);
- 13. Any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the patient or the quality of study data;
- 14. Planned or prior participation in any other interventional drug study within 30

### Study Procedures

### Screening/Baseline

Screening/Baseline assessments and procedures must be completed within 24 hours before the start of the study drug infusion. Potential subjects who do not meet enrollment criteria may, as appropriate, repeat the screening assessments once at a later time for possible enrollment into the study. Local laboratory results will be used to determine subject eligibility for study enrollment. Any protocol-required eligibility laboratory evaluations already done as part of the patient's regular medical care within 24 hours before the start of the study drug infusion on Study Day 1 do not have to be repeated for purposes of determining eligibility for this study.

- Obtain informed consent in writing from patient, legal authorized representative, or next of kin, according to local regulations.
- Clinical Assessments:
  - Obtain a complete medical and surgical history, including: a) all active conditions and all conditions diagnosed within the previous 1 year
  - Perform a complete physical examination (general/appearance; head, eyes, ears, nose, and throat [HEENT]; neurological; pulmonary; cardiovascular; gastrointestinal; musculoskeletal; and skin)
  - Record height and weight
  - Record resting pulse, blood pressure, and respiratory rate; oxygen saturation (by pulse oximeter), including rate of supplemental oxygen (i.e., FiO2); ventilator support; and highest (or lowest if hypothermia) daily temperature (oral, rectal, tympanic, or core) measured
  - Record total fluid balance including total fluid intake and total fluid output for the period encompassing the signing of the ICF to the start of the study drug infusion
  - Record each component of the Acute Physiology and Chronic Health Evaluation II (APACHE II) assessment at Screening/Baseline

MISP Template: Protocol Final Version: 8/13/2010

- Record all prior medications taken or received within 3 days before study drug infusion
- Identify, assess, and record any new adverse events or Serious Adverse Events (SAE) after signing of informed consent
- Laboratory Assessments:
  - Collect the following labs within 24 hours of study dose administration: serum creatinine, blood urea nitrogen, glucose, sodium, potassium, chloride, bicarbonate, albumin, total protein, complete blood count (CBC) with differential, total bilirubin, direct bilirubin, alkaline phosphate, alanine aminotransferase, aspartame aminotransferase, and urine analysis with microscopy. A serum hCG test will be collected for females of child-bearing potential.
  - Calculation of CrCL using Cockcroft-Gault based on screening/baseline serum creatinine:

Calculated CrCL =  $(140 - age in years) \times ideal body weight (kg)^{a,b,c}$  $72 \times SCr (mg/dL)$ 

### Multiply by 0.85 for female patients

- a Ideal body weight (IBW, kg): Males = 50 + [2.3 × (Height (in) 60)]; Females = 45.5 + [2.3 × (Height (in) - 60)]
- b For patients with total body weight (TBW) that is greater than 20% over IBW, use adjusted body weight (ABW, kg): IBW + 0.4\*(TBW-IBW)
- <sup>c</sup> If TBW is less than IBW, use TBW in equation

### Study Medication Administration

All participants will receive a single dose of imipenem-cilastatin-relebactam 1.25 grams as a 30 minute (+/- 5 minutes) infusion. Imipenem-cilastatin-relebactam vials will be supplied by the study sponsor. The dose will be prepared according to manufacturer recommendations in precisely 100 ml of 0.9% sodium chloride. Imipenem-cilastatin-relebactam must be administered through a peripheral intravenous catheter, peripherally inserted central catheter (PICC), central line, or port-a-catheter, whichever is determined to be most appropriate by the local investigator and care provider for each participant. Participants will also receive standard intravenous antibiotic therapy (excluding generic or branded intravenous imipenem) to treat their suspected infection, as determined by the responsible provider. No other intravenous medications will be co-administered with imipenem-cilastatin-relebactam.

### Study Day 1

- Within 8 hours of beginning study medication infusion, a pre-dose SCr will be collected to confirm calculated CrCL remains ≥130 mL/min and that no change in SCr was observed to be ≥ 0.3 mg/dL from the baseline SCr used qualifying for enrollment.
- An 8 hour (± 1 hour) urine creatinine collection will be initiated within 4 hours prior to study medication infusion. The results of the measured urine CrCL will be used to confirm ARC in the patient over the time period that blood samples for imipenem-cilastatin-relebactam are collected.

MISP Template: Protocol 6 Final Version: 8/13/2010

### Measured CrCL (ml/min) = UCr (mg/dL) x urine volume (mL) Predose-SCr x timea

Abbreviations: CrCl = creatinine clearance; SCr = serum creatinine; UCr = urine creatinine.

- <sup>a</sup> Time = The 8-hour urine collection has a ± 1 hour window (i.e., 480 min ± 60 min); use the exact number of minutes of the urine collection in the equation
- Vital signs (temperature, heart rate, blood pressure, respiratory rate) will be recorded within 15 minutes prior to starting the study drug infusion.
- Participants will receive the single dose of imipenem-relebactam as described above. Exact start and stop times will be recorded in military time.
- Identify, assess, and record any new adverse events or Serious Adverse Events (SAE)
- Concomitant medications will be recorded.
- Blood Sample Collection: Seven blood samples (4 ml per sample) will be collected in K2EDTA vacutainers at the following time points to determine the concentrations of imipenem and relebactam in plasma: 0 hour (within 30 minutes prior to the start of infusion), 0.5 hours (end of infusion), 0.75, 1, 2, 4, and 6 hours after the start of the infusion. The timing of all blood samples should be +/- 5 minutes of protocol defined time, except for the 0.5 hour (peak concentration), which can be + 5 minutes and should be collected as close to the end of the infusion as possible. All blood samples will be collected via a peripheral intravenous catheter inserted into the contralateral arm to drug administration for collection of blood samples. Alternatively, venipuncture may be used to collect the seven blood samples.
- Blood samples will be immediately stored on ice and centrifuged within 30 minutes of collection at 1000-1300 x g (rcf) for 10 minutes at 4°C to separate the plasma.
- Immediately after centrifugation of whole blood, use a 1.0 mL pipette to transfer exactly 1.0 mL of plasma to labeled, cryovials containing 1.0 mL of plasma stabilizer (2-(N-morpholino) ethanesulfonic acid (MES)). Add a second 1.0 mL of plasma to a second cryovial to serve as a back-up sample.
- Cap the cryovials and mix the plasma with the preservative stabilizer by inverting at least six times. Freeze and store at -80 °C. No more than 60 minutes should elapse between the blood draw and freezing of plasma
- An additional 8ml blood sample will be collected for imipenem and relebactam protein binding determination at 0.5 hours (end of infusion). Plasma will be separated by centrifugation as previously explained. Approximately 0.9 mL of plasma will be loaded in an ultrafiltration device (Centrifree®, Merck Millipore Ltd., Ireland) and centrifuged for 45 minutes at 10° C at 2,000 x g to obtain an ultrafiltrate containing only free-drug concentrations. Protein binding will be conducted in triplicate. The proteinfree ultrafiltrate volume will be measured, transferred to a cryovial and then, an equal volume of the stabilizer will be added (confirmation of processing instructions for protein-free imipenem and relebactam will be provided by Q2 Solutions, Ithaca, NY). The cryovials will be stored at -80° C until concentration determination. The final protein percentage will be calculated by dividing the free concentration by the total plasma concentration and subtracting from 100 (%).

### Study Day 2

- Clinical Assessments:
  - Perform a complete physical examination

# Record resting pulse, blood pressure, and respiratory rate; oxygen saturation (by pulse oximeter), including rate of supplemental oxygen (i.e., FiO2); ventilator support; and highest (or lowest if hypothermia) daily temperature (oral, rectal, tympanic, or core) measured Identify, assess, and record any new adverse events or Serious Adverse Events (SAE) Laboratory Assessments:

 Collect the following labs within 24 hours after completion of last blood sample collection: serum creatinine, blood urea nitrogen, glucose, sodium, potassium, chloride, bicarbonate, albumin, total protein, complete blood count (CBC) with differential, total bilirubin, direct bilirubin, alkaline phosphate, alanine aminotransferase, aspartame aminotransferase, and urine analysis with microscopy.

## 2.6 Study Duration

Final Protocol 2 months
IRB Approval 2 months
Enrollment and Sampling 10 months
Imipenem-relebactam Analytical (by Sponsor) TBD
Pharmacokinetic Analyses 1 months
Final Report 1 months

### **Data Analyses**

### Data Collection

Patient demographics, medical/surgical history, concomitant medications, and adverse event data will be collected throughout the study on a provided case report form. Protected Health Information (PHI) will be maintained at CAIRD.

### Analysis Populations

All patients enrolled will be included in the safety population. However, only the 8 patients who meet the definition of ARC will served as the primary pharmacokinetic population. Any additional patients enrolled who do not meet the definition of ARC will have imipenem and relebactam concentrations determined for informational purposes. These patients will not be included in the summary pharmacokinetic analyses.

### 2.7 Statistical Analysis and Sample Size Justification

### Analytical

Cryovials containing plasma and protein free filtrate will be overnight shipped on dry ice to Q2 Solutions (Ithaca, NY) for imipenem and relebactam concentration determination. The back-up vial will be shipped separately. Imipenem and relebactam concentrations will be determined by a liquid chromatography mass spectrometry assay.

### Pharmacokinetic Analyses

### Non-compartmental

Non-compartmental modeling will be conducted using WinNonlin (Pharsight Corporation, Cary, NC) using the latest version licensed for the laboratory. All concentration time curves will be plotted for visual inspection. The following pharmacokinetic parameters will be estimated for imipenem and relebactam in each of the 8 participants. The maximum concentration ( $C_{max}$ ) will be the highest concentration observed for the concentration time profile of each participant. The time to maximum concentration ( $T_{max}$ ) will be the observed sampling time of the  $T_{max}$ . The minimum concentration ( $T_{min}$ ) will be the lowest concentration observed for the concentration time profile of each participant that occurs after the observed  $T_{max}$ . Lambda ( $T_{max}$ ) will be the resulting slope of the regression line

MISP Template: Protocol 8 Final Version: 8/13/2010

of best fit. Half-life  $(T_{1/2})$  will be calculated as  $\ln(2)/\lambda_z$ . Area under the curve for the dosing interval  $(AUC_{0-\tau})$  will be calculated by the linear/log trapezoidal rule (linear during increasing concentrations, log during decreasing concentrations), where  $\tau$  is the dosing interval for the drug studied. The AUC to infinity  $(AUC_{INF})$  will be calculated as the AUC extrapolated to infinity by the equation: AUC +  $C_{last}/\lambda_z$ . Clearance (CL) will be estimated by Dose/AUC $_{0-\tau}$ . The volume of distribution based on the terminal elimination phase  $(V_z)$  will be estimated by Dose/ $(\lambda_z^*AUC_{0-\tau})$ .

### Population Pharmacokinetic Analyses

Imipenem and relebactam concentrations will be modeled using the non-parametric adaptive grid program (NPAG) with adaptive gamma in the Pmetrics package for R (Laboratory of Applied Pharmacokinetics and Bioinformatics, Los Angeles, CA) using either a one or two compartment model. Appropriate model selection will be based on visual inspection, observed versus predicted plots, and Akaike Information Criterion (AIC). The effect of specific body size descriptors (actual body weight, ideal body weight, body mass index, body surface area) and both calculated and measured CrCL will be analyzed for correlation with pharmacokinetic parameters (i.e., CL and volume of distribution).

### Monte Carlo Simulation

Using the population pharmacokinetic model, a 5000 patient Monte Carlo simulation will be conducted for the standard imipenem and relebactam dosing regimen to determine probability of achieving pharmacodynamic thresholds, as defined by Sponsor, at the imipenem susceptibility breakpoint of 2  $\mu$ g/mL. Observed fraction unbound estimates from the protein-free ultrafiltrate studies in these patients will be incorporated into simulations. In the scenario that the probability of target attainment (PTA) is less than 90%, a higher dose and longer infusion time (e.g., 2-3 hours) will be simulated to determine a dose that achieves at least 90% PTA. Analyses will also be conducted using contemporary MIC distributions of *P. aeruginosa* and KPC producing *K. pneumoniae*.

### Power/Sample Size:

Based upon relebactam single dose pharmacokinetic data from healthy volunteers receiving the drug with or without imipenem (3), clearance across all doses was 8.6 L/h with a standard deviation of 1.2 L/h. Eight in the ARC group would provide 80% power at an alpha of 0.05 to detect a 40% difference in total body clearance from the historical healthy volunteer data; this also assumes an increase in coefficient of variability (CV) to 25%, which is expected in critically ill patients. Since some patients with calculated CrCL via Cockcroft-Gault will not have 8 hour urine CrCL of at least 130 ml/min/1.73 m², this study will enroll up to 12 patients to have complete data for 8 patients with ARC. Enrollment will stop once complete data for 8 patients who meet the definition of ARC is confirmed or a maximum of 12 patients complete the study, whichever occurs first.

### 2.8 Specific Drug Supply Requirements

Imipenem-Cilastatin-Relebactam 1.25 gram vials (n=15 vials)

### Participants will be monitored for any sign or symptom of adverse events throughout the course of the study. Unanticipated, life-threatening or fatal adverse events will be reported to the IRB, the manufacturer, and the Food and Drug Administration according to federal guidelines. All adverse events requiring medical attention will be treated by the study physician and will be recorded by the investigator.

For the purpose of this study, an adverse event will be defined as any pathologic or unintended change in the structure (signs), function (symptoms), or chemistry (laboratory values) of the body associated with the use of the study drug, whether or not considered drug related, and will be categorized as one of the following:

- MILD present, but easily tolerated
- MODERATE discomfort that interferes with usual activities
- SEVERE incapacitating, inability to work or do usual activities

### 2.9 Adverse Experience Reporting

Relationship of the AE to the study medication (i.e., causality) will be evaluated according to the investigator's opinion, as one of the following:

- Concurrent condition unrelated to study drug
- REMOTE adverse drug event little or no temporal relationship to study
- POSSIBLE adverse drug event temporal relationship to study drug
- PROBABLE adverse drug event commonly associated with study drug
- DEFINTE adverse drug event reappeared on re-challenge of study drug

All SAEs will be reported to the Institutional Review Board, sponsor, and the Food and Drug Administration according to Federal and local guidelines. A serious adverse event will be defined as any adverse event that results in death, is immediately life-threatening, requires or prolongs hospitalization, or is an important medical event that may jeopardize the participant or may require medical intervention to prevent one of the previously mentioned outcomes.

### 2.10 Itemized Study **Budget**

### See Proposed Budget

### 2.11 References

- Zhanel GC, Lawrence CK, Adam H, Schweizer F, Zelenitsky S, Zhanel M, Lagace-wiens PRS, Walkty A, Denisuik A, Golden A, Gin AS, Hoban DJ, Lynch JP, Karlowsky JA. Imipenem-relebactam and meropenemvaborbactam: two novel carbapenem-beta-lactamase inhibitor combinations. Drugs 2018:78:65-98.
- 2. Lob SH, Hackel MA, Kazmierczak KM, Young K, Motyl MR, Karlowsky JA, Sahm DF. In vitro activity of imipenem-relebactam against gram-negative ESKAPE pathogens isolated by clinical laboratories in the United states in 2015 (results from the SMART global surveillance program). Antimicrob Agents Chemother 2017;61:e02209-16.
- 3. Rhee EG, Rizk ML, Calder N, Nefliu M, Warrington SJ, Schwartz MS, Mangin E, Boundy K, Bhagunde P, Colon-Gonzalez F, Jumes P, Liu Y, Butterton JR. Pharmacokinetcs, safety, and tolerability of single and multiple doses of relebactam, a beta-lactamase inhibitor, in combination with imipenem and cilastatin in healthy participants. Antimicrob Agents Chemother 2018;62:e00280.
- 4. Udy AA, Roberts JA, Shorr AF, Boots RJ, Lipman J. Augmented renal clearance in septic and traumatized patients with normal plasma creatinine

MISP Template: Protocol Final Version: 8/13/2010

IRB NUMBER: HHC-2019-0237 IRB APPROVAL DATE: 12/22/2020

| | concentrations: identifying at-risk patients. Crit Care 2013;17:R35. 5. Udy AA, Baptista JP, Lim NL, Joynt GM, Jarrett P, Wockner L, Boots RJ, Lipman J. Augmented renal clearance in the ICU: results of a multicenter observational study of renal function in critically ill patients with normal plasma creatinine concentrations. Crit Care Med 2014;42:520-7. 6. Troger U, Drust A, Martens-Lobenhoffer J, Tanev I, Braun-Dullaeus RC, Bode-Boger SM. Decreased meropenem levels in intensive care unit |
|---|---|
| | patients with augmented renal clearance: benefit of therapeutic drug monitoring. Int J Antimicrob Agents 2012;40:370-2. 7. Carler M, Carrette S, Roberts JA, Stove V, Verstraete A, Hoste E, Depuydt P, Decruyenaere J, Lipman J, Wallis SC, De Waele JJ. Meropenem and piperacillin/tazobactam prescribing in critically ill patients: does augmented renal clearance affect pharmacokinetic/pharmacodynamic target attainment when extended infusions are used? Crit Care 2013;17:R84. |
| | <ol> <li>De Waele JJ, Lipman J, Akova M, Bassetti M, Dimopoulos G, Kaukonen M, Koulenti D, Martin C, Montravers P, Rello J, Rhodes A, Udy AA, Starr T, Wallis SC, Roberts JA. Risk factors for target non-attainment during empirical treatment with β-lactam antibiotics in critically ill patients. Intensive Care Med 2014;40:1340-51.</li> </ol> |
| | 9. Huttner A, Von Dach E, Renzoni A, Huttner BD, Affaticati M, Pagani L, Daali Y, Pugin J, Karmime A, Fathi M, Lew D, Harbarth S. Augmented renal clearance, low β-lactam concentrations and clinical outcomes in the critically ill: an observational prospective cohort study. Int J Antimicrob Agents 2015;45:385-92. |
| | 10. Bergen PJ, Bulitta JB, Kirkpatrick CMJ, Rogers KE, McGregor MJ, Wallis SC, Paterson DL, Nation RL, Lipman J, Roberts JA, Landersdorfer CB. Substantial impact of altered pharmacokinetics in critically ill patients on the antibacterial effects of meropenem evaluated via the dynamic hollow-fiber infection model. Antimicrob Agents Chemother 2017;61:e02642-16. |
| 2.12 Publication<br>Plan | The results of this study would be presented at an international congress such as the ASM Microbe Meeting, IDWeek, ECCMID, or SCCM. A final publication would be submitted to a peer reviewed journal such as Antimicrobial Agents and Chemotherapy or Journal of Antimicrobial Chemotherapy. |
| 2.13 Curriculum<br>Vitae | Investigator should provide curriculum vitae in English and a listing of references to MSD. |
| 2.13 Protocol<br>Submission for<br>Investigator- | U.S. protocols should be submitted by US investigators directly or through the Global Research Specialist at <a href="https://www.merckiisp.com">www.merckiisp.com</a> |
| Initiated Studies | Non U.S. protocols should be submitted to the MSD office by the investigators. |